CLINICAL TRIAL: NCT00502411
Title: A Phase I Study of Post-Operative Concurrent Chemoradiation for Extremity and Trunk Soft Tissue Sarcoma
Brief Title: Post-Operative Chemoradiation for Extremity & Trunk Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-336; NCI-2012-01519 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft Tissue Sarcoma; External Beam Radiotherapy; Radiation Therapy; Extremity and Trunk; EBRT; Sarcoma; Doxorubicin; AD; Hydroxydaunomycin hydrochloride; XRT; RT; Radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxorubicin + Radiation Therapy (Experimental): Doxorubicin 17.5 mg/m^2 IV bolus infusion, followed by continuous IV infusion on days 1-4. Radiation treatments 5 days a week for 6 - 6 1/2 weeks. 60 Gy in 6 weeks (negative resection margin) to 66 Gy in 6.5 weeks (positive resection margin).
  Interventions: Drug: Doxorubicin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Doxorubicin — 17.5 mg/m^2 IV bolus infusion, followed by continuous IV infusion on days 1-4.
  Other Names: AD; Hydroxydaunomycin hydrochloride
Radiation: Radiation Therapy — Radiation treatments 5 days a week for 6 - 6 1/2 weeks. 60 Gy in 6 weeks (negative resection margin) to 66 Gy in 6.5 weeks (positive resection margin).
  Other Names: XRT; RT; Radiotherapy

SUMMARY:
The goal of this clinical research study is to learn if the combination of radiation therapy plus low dose doxorubicin chemotherapy given after surgery is effective in the treatment of sarcoma. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Doxorubicin is a drug that is commonly used to treat certain kinds of cancer.

The radiation treatment and chemotherapy will start around 4-6 weeks after surgery. During the study, you will receive radiation treatments 5 days a week for 6 - 61/2 weeks. On Day 1 of each week of radiation therapy, you will be given doxorubicin through a continuous injection into a vein for 4 days in a row. A special tube is placed into a large vein in the neck or chest region or through a large vein in the arm. This is called a central venous line. A small pump is then used to give the drug. This pump is about the size of a pack of cigarettes. You will receive appropriate instructions for the maintenance of the pump. The doxorubicin and radiotherapy will be given on an outpatient basis at M. D. Anderson.

If the disease gets worse or you experience any intolerable side effects, chemotherapy and/or radiation therapy may be stopped and you may be taken off the study. At that time, your doctor will discuss other treatment options with you.

Before the start of each week of treatment, you will have a physical exam and blood tests (around 2 tablespoons). You will also have a MRI to check on the status of the disease.

After the study, you will have follow-up visits at M. D. Anderson every 3-4 months for the first 2 years after the study then every 6 months for the next 3 years. After that you will have follow-up visits once a year for the rest of your life to check on the status of the disease. At every follow-up visit you will have ultrasound scans. You will have a MRI at the first follow-up visit then only when the doctor feels it is necessary.

This is an investigational study. Doxorubicin is FDA approved and is commercially available. Up to 30 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with cytological or histological proof of large (> 5 cm), completely resected soft tissue sarcoma of the extremity or trunk (AJCC Stage IB, IIA, IIC, and III) will be eligible. Patients with stage IV sarcoma who are considered for primary tumor treatment with surgery and postoperative radiation are also eligible.
2. Patients who have undergone pre-referral surgical resection or excisional biopsy with no measurable residual disease on appropriate radiological imaging will be eligible. The adequacy of the surgical resection will be evaluated at MDACC and re-excision will be performed as necessary. Negative surgical resection margins are desirable; positive margins, however, are allowable if re-excision would result in functional deficit.
3. Patients may have received prior doxorubicin-based systemic chemotherapy up to a total doxorubicin dose of 450 mg/m2. Inclusion of patients with a prior history of malignancy will be at the discretion of the Study Chairman.
4. Patients must have a Karnofsky P.S. of > 70 or a Zubrod P.S. of 0 or 1.
5. Absolute neutrophil count must be > 1,500 cells/mm; platelet count > 100,000 platelets/ml; serum creatinine < 1.8 mg/dl, serum glutamate oxaloacetate transaminase (SGOT)/serum glutamate pyruvate transaminase (SGPT) < 3 x normal, total bilirubin < 1.5 mg/dl. For patients with cumulative doxorubicin 400 - 450 mg/m2, EF > 50%.
6. EKG (within 6 weeks of the planned start of treatment).
7. Echocardiogram or multiple gated acquisition scan (MUGA) (if prior doxorubicin treatment or history of either myocardial infarction or congestive heart failure).
8. Patients must have no uncontrolled co-existing medical conditions.
9. Women of childbearing potential must not be pregnant or breast feeding and must practice adequate contraception.
10. All patients must sign an informed consent.

Exclusion Criteria:

1) Patients with a history of prior radiotherapy in the area of the primary tumor or those in whom the anticipated radiation field would include the perineum, scrotum, or vaginal introitus will not be eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Toxicity of Radiation Therapy Plus Low Dose Doxorubicin in Participants with Extremity and Trunk Sarcoma | 6 weeks after the start of Doxorubicin
  Toxicity defined by acute local toxicity to skin and subcutaneous tissues and delayed wound healing. Toxicity defined as (1) grade 3 or 4 myelosuppression with fever or (2) grade 3 or 4 desquamation, or (3) both (1) and (2), scored within 6 weeks from the start of doxorubicin treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Pisters, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org